CLINICAL TRIAL: NCT01934647
Title: A Non-randomized, Single-Panel, Open-Label Trial to Study the Safety, Tolerability and Pharmacodynamics of MK-8892 Acute Dosing in Subjects With Moderate to Severe Pulmonary Arterial Hypertension
Brief Title: Acute Dosing of MK-8892 in Participants With Pulmonary Arterial Hypertension (PAH) (MK-8892-003)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8892-003; 2013-001680-23 (EudraCT Number); MK-8892-003 (Other: Merck Protocol Number)
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 mg MK-8892 (Experimental): Participants will receive a single oral dose of 1 mg MK-8892.
  Interventions: Drug: MK-8892
- 4 mg MK-8892 (Experimental): Participants will receive a single oral dose of 4 mg MK-8892.
  Interventions: Drug: MK-8892
- 8 mg MK-8892 (Experimental): Participants will receive a single oral dose of 8 mg MK-8892.
  Interventions: Drug: MK-8892

INTERVENTIONS:
Drug: MK-8892 — Single oral capsule with 1 mg, 4 mg, or 8 mg of MK-8892

SUMMARY:
This clinical trial will study the safety, tolerability, and pharmacodynamics of single doses of MK-8892 in participants with pulmonary arterial hypertension (PAH). The primary objective is to estimate the measured peak effect of the highest acutely tolerated (HAT) single oral dose of MK-8892 on pulmonary vascular resistance (PVR).

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal female or if female of reproductive potential, remains abstinent or uses two acceptable methods of birth control during 14 days after dosing with MK-8892
* has suspected PAH classified in one of the following sub-groups: idiopathic, heritable, drug- or toxin-induced, or associated with connective tissue disease, as defined by the Dana Point 2008 Clinical Classification
* has a clinical indication for right heart catheterization
* PAH classified as World Health Organization (WHO) functional class II or III

Exclusion Criteria:

* has a medical history indicating a secondary cause of Pulmonary Hypertension (PH) or a non-included etiology of PAH including the following tests within 6 months of Visit 1: Echo indicating significant left heart disease, valvular disease, or structural defects; function test indicating significant pulmonary disease; imaging test indicating veno-occlusive disease; perfusion scan indicating thromboembolic disease; abdominal ultrasound indicating cirrhosis; positive test for human immunodeficiency virus (HIV)
* has persistent or permanent atrial fibrillation, significantly impaired gas exchange, history of radiation of the lung or mediastinum, hepatic or hepatobiliary disease, immunodeficiencies or latent bleeding risk
* has estimated Glomerular Filtration Rate (GFR) <45 mL/min
* has alanine aminotransferase test (ALT) serum glutamic pyruvic transaminase (SGPT) or aspartate aminotransferase test (AST) serum glutamic oxaloacetic transaminase (SGOT) >= 3 x upper limit of normal (ULN) at Visit 1
* has a systolic blood pressure (BP) <105 mmHg, or heart rate (HR) > 100 beats/min at Visit 1 (Day -7 to -1)
* has previously received specific therapy for PAH within 4 weeks prior to Visit 1
* has taken sildenafil, valdenafil or a nitrate within 24 hours prior to Visit 2 date
* has taken tadalafil within 7 days prior to Visit 2 date
* has taken 2 or more specific PAH medications concomitantly within 4 weeks of anticipated Visit 2 date. Only treatment naïve subjects or subjects on stable PAH-specific monotherapy with an endothelin receptor antagonist ([ERA]; bosentan, ambrisentan, or macitentan) or a prostacyclin analog ([PCA]; treprostinil, epoprostenol, or iloprost) are eligible. PAH monotherapy with one of these medications may continue without interruption during this study
* has taken a soluble guanylate cyclase (sGC) activator (riociguat) within 24 hours of anticipated Visit 2 date.
* has taken diltiazem immediate release within 1 day or diltiazem extended release within 2 days prior to Visit 2 date
* is currently taking potent inhibitors or inducers of Cytochrome P450 3A4 (CYPA4), or is consuming >1 liter of grapefruit juice per day
* is pregnant or breastfeeding or expecting to conceive during study or post study follow-up period
* has donated 500 mL of blood within prior 60 days
* is currently participating in or has within the prior three months participated in a study with an investigational compound or device

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-11-22 (Actual); Primary Completion 2014-09-08 (Actual); Study Completion 2014-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 mg MK-8892: Participants received a single oral dose of 1 mg MK-8892.
- 4 mg MK-8892: Participants received a single oral dose of 4 mg MK-8892.
- 8 mg MK-8892: Participants received a single oral dose of 8 mg MK-8892.
Period: Overall Study
Arm/Group | 1 mg MK-8892 | 4 mg MK-8892 | 8 mg MK-8892
Started | 2 | 2 | 3
Completed | 2 | 2 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mg MK-8892 | 4 mg MK-8892 | 8 mg MK-8892 | Total
Number analyzed (Participants) | 2 | 2 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.5 (17.7) | 52.0 (1.4) | 61.3 (11.0) | 51 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 0 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Peak Percent Change From Baseline in Pulmonary Vascular Resistance (PVR) at the Highest Acutely Tolerated (HAT) Dose of MK-8892
Description: PVR assessments were performed throughout the right heart catheterization (RHC). Peak PVR reduction was determined to occur if 2 consecutive PVR measurements were at least 20% greater than the nadir PVR measurement.
Time Frame: Baseline and up to 5 hours post-dose
Population: Planned efficacy analysis could not be performed due to early study termination.
Arm/Group | 1 mg MK-8892 | 4 mg MK-8892 | 8 mg MK-8892
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 14 days after study drug administration
Description: Safety analysis included all participants who received at least one dose of study drug.
Groups:
- Panel A: 1 mg: Participants received a single oral dose of 1 mg MK-8892.
- Panel B: 4 mg: Participants received a single oral dose of 4 mg MK-8892.
- Panel C: 8 mg: Participants received a single oral dose of 8 mg MK-8892.
Arm/Group | Panel A: 1 mg | Panel B: 4 mg | Panel C: 8 mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: 1 mg (N=2) | Panel B: 4 mg (N=2) | Panel C: 8 mg (N=3)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.